CLINICAL TRIAL: NCT04686162
Title: Bae: A Smartphone Application for a Better Following Adolescents at Risk of Suicidal
Brief Title: Bae: A Smartphone Application for a Better Following Adolescents at Risk of Suicidal Behavior: Study of Acceptability and Preliminary Results of Efficacy
Acronym: BAE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: University Hospital, Lille (Other); University Hospital, Nîmes (Unknown); La Timone Hospital, Marseille (Unknown); Association "Mal être des adolescents", Marseille (Unknown); Salvator Hospital, Marseille (Unknown); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Laboratoire d'Informatique, de Robotique et de Microélectronique de Montpellier (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RECHMPL20-0153; 2020-A03150-39 (Other: ANSM)
Record Dates: First submitted 2020-12-22; First posted 2020-12-28 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-02

CONDITIONS: Suicide Attempt; Suicidal Ideation
Keywords: suicide attempt; suicidal ideation; e-Health; smartphone application; ecological momentary assessment; adolescents
MeSH Terms: conditions — Suicide, Attempted; Suicidal Ideation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group using the smartphone application bae (Experimental): Patients with personal history of suicide attempt or with suicidal ideation, will use the application during 6 months.
  Interventions: Other: bae application

INTERVENTIONS:
Other: bae application — Patients will be assisted by a research team member to install and configure the application bae on their smartphone; then, they will be trained to use it.
  Bae proposes 4 types of assessments :
  1. 5 times a day during 3 days, every month (5 minutes) : patients can assess their emotions, their thoughts, their behavior and their occurrence context.
  2. Weekly (7 minutes) : consists of a summary of the week, about their emotions, thoughts, behavior, their relationships (family, work, friends), and their quality of life.
  3. Monthly (5 minutes): assessment of the usefulness and satisfaction about the application.
  4. Assessment available at any time An action plan is designed to support the participants, to help them facing difficult emotions and feelings, and to encourage them to ask for help.
  They can contact a relative or call the psychiatric emergency service directly by clicking on a button.
  Patients can try to identify their own warning signs, to prevent suicidal behavior.

SUMMARY:
Suicidal behavior among adolescents is a major public health problem. Exacerbation of suicidal risk most often occurs when the young person is in his or her natural environment, far from the health care system. Therefore, real-time risk detection would make it possible to deploy immediate action interventions. A smartphone application for personalized assessment and intervention would enable patients to better anticipate and manage suicidal crises and stay connected to the healthcare system. The increasing use of smartphones and mobile applications among adolescents supports the feasibility and value of such follow-up among young people. In a first phase of this project, investigators first undertook to develop bae: a smartphone application adapted to a population of adolescents collecting information on their suicidal behaviour in a contextualized manner, with the added benefit of offering emotion management modules as well as personalized psychoeducational messages and alerts delivered to young people in the event of a crisis. The application is intended to be a complementary tool to the usual treatment. Before testing its effectiveness and due to the novelty of the intervention, a rigorous feasibility study in a real clinical context is necessary to ensure acceptability and satisfaction with the use of the bae application.

The objective is to evaluate, over a 6-month period, the acceptability of a follow-up of a population of 100 adolescents (12-17 years) at risk of suicidal driving via the bae smartphone application.

DETAILED DESCRIPTION:
100 patients having recently attempted suicide or having suicidal ideation will be recruited. They will be asked to use the application bae during 6 months and will be followed up during this period.

Initial visit (inclusion) : clinical assessment and installation of the application bae.

Last visit (6th month) : clinical assessment.

ELIGIBILITY:
Criteria for inclusion

All subjects will be required to meet the following inclusion criteria:

* Having consulted in the context of a suicidal crisis according to the criteria defined according to the consensus conference of the High Authority of Health (HAS 2000) ("psychic crisis for which the major risk is suicide. It can be represented as the trajectory that goes from the pejorative feeling of being in a situation of failure to a perceived impossibility of escaping this impasse. It is accompanied by suicidal ideas that become more and more pervasive and pervasive until the eventual act is carried out") in the previous 7 days.
* Possess a compatible smartphone (operating system: iOs or Androïd)
* Subject affiliated to or beneficiary of a French social security scheme
* Be able to understand the nature, purpose and methodology of the study
* Informed consent signed by the patient and his/her parent(s) or legal representative(s)

Exclusion Criteria:

* Patient deprived of liberty (by judicial or administrative decision)
* Inability to understand, speak and write French
* Participation in another study with an exclusion period.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2021-09-20 (Estimated); Primary Completion 2022-07-11 (Estimated); Study Completion 2022-07-11 (Estimated)

PRIMARY OUTCOMES:
Acceptability | at 6 months
  Rate of completion of the ecological momentary assessment questionnaires.

SECONDARY OUTCOMES:
Prevention modules use | 6 months
  The number of times the patient uses prevention modules
Call module use | 6 months
  The number of calls made through the application to relatives/psychiatry/samu services
Satisfation | 1, 2, 3, 4, 5 and 6 months
  Satisfaction is assessed by monthly questionnaires in the application (Likert scales from 0 to 10, 0 is the worst and 10 the best)
Satisfaction | 6 months
  Satisfaction is assessed by a self administrated questionnaire to be completed during the telephone interview at 6 months by a Likert scales from 0 to 10, 0 is the worst and 10 the best)
Occurrence of a suicidal event | 6 months
  The occurrence of a suicidal event will be assessed by The Columbia-Suicide Severity Rating Scale